CLINICAL TRIAL: NCT03279861
Title: Sacubitril-valsartan (Entresto) Versus Standard Anti-hypertensive Therapy in LVAD Patients - A Feasibility Pilot Study
Brief Title: Sacubitril-valsartan Versus Usual Anti-hypertensives in LVAD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: protocol change
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00076889
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2018-02

CONDITIONS: Congestive Heart Failure; Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entresto (Active Comparator): First-line anti-hypertensive: sacubitril-valsartan, starting at 24-26 mg twice daily, increasing to maximum dose of 97-103 mg twice daily
  Interventions: Drug: Entresto; Drug: Valsartan
- Usual meds (Active Comparator): First-line anti-hypertensive: valsartan, starting at 40 mg twice daily, increasing to a maximum dose of 160 mg twice daily
  Interventions: Drug: Entresto; Drug: Valsartan

INTERVENTIONS:
Drug: Entresto — First line therapy in Entresto arm
Drug: Valsartan — First line therapy in "usual meds" arm

SUMMARY:
This pilot, feasibility study evaluates the efficacy of sacubitril-valsartan (Entresto) versus usual anti-hypertensive medications in patients with left ventricular assist devices (LVAD). It also measures diurnal blood pressure variations in the context of continuous flow physiology.

DETAILED DESCRIPTION:
Left ventricular assist devices (LVAD) have become a life-saving therapy for patients with ACC/AHA stage D congestive heart failure (CHF). Despite longevity and improved quality of life, LVAD-supported patients are plagued with adverse events, the most debilitating of all is stroke. Ischemic and hemorrhagic strokes have been associated with hypertension (mean arterial pressure, or MAP > 90 mmHg) in addition to out-of-range INR and aspirin doses. Strict blood pressure control has been shown in a recent randomized trial to confer a significant decline in stroke rates of patients implanted with the Heartware LVAD. Patients with poorly controlled hypertension are also at risk for inadequate left-ventricular unloading and worsening CHF due to the exquisite sensitivity to afterload of the continuous flow LVAD.

There are no guidelines for the use of anti-hypertensives in LVAD patients. Most are started on standard CHF therapies, though this practice varies greatly across LVAD centers. The angiotensin receptor blocker-neprilysin inhibitor sacubitril-valsartan (Entresto) is a potent anti-hypertensive mediation that was recently approved by the Food and Drug Administration for the treatment of patients with heart failure and low ejection fraction. We aim to randomly assign patients to receive Entresto or usual anti-hypertensive therapy for blood pressure control, then crossover to the other arm after 30 days. Daily blood pressure measurements will be performed and correlated with LVAD pump flows and waveform analysis.

ELIGIBILITY:
Inclusion Criteria:

* More than 30 days after LVAD implant
* Ambulatory
* MAP > 85 mmHg requiring initiation of anti-hypertensive medications

Exclusion Criteria:

* Allergy to ACEI or ARB
* eGFR < 30 mL/min/1.73m2
* K > 5.4 mmol/L
* MAP < 60
* Inability to check blood pressure at home
* Lack of prescription coverage
* Frequent hospitalizations (monthly)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Time spent with MAP < 85 mmHg | 2 months
  Daily mean arterial pressure (MAP) < 85 mmHg

SECONDARY OUTCOMES:
Number of drugs | 2 months
  Number of anti-hypertensive drugs needed to achieve MAP < 85 mmHg
Pump flow | 2 months
  Correlation of pump flow with daily MAP

CONTACTS AND LOCATIONS:
Overall Officials: Van-Khue Ton, MD PhD, Principal Investigator — University of Maryland

IPD SHARING:
Plan to Share IPD: No